CLINICAL TRIAL: NCT00151788
Title: A Randomized, Double-blind, Stratified, Placebo-controlled, Parallel-group Study of the Efficacy and Safety of the ACAT Inhibitor CS-505 for Reducing the Progression of Atherosclerosis in Subjects With Heterozygous Familial Hypercholesterolemia and Carotid Atherosclerosis Using Carotid Ultrasound (CUS)
Brief Title: Efficacy and Safety of the ACAT Inhibitor CS-505 (Pactimibe) for Reducing the Progression of Carotid Artery Disease. This Study is Also Known as CAPTIVATE.
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 505-205
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Atherosclerosis; Heterozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Atherosclerosis | interventions — pactimibe

INTERVENTIONS:
Drug: Pactimibe sulfate

SUMMARY:
The effects of pactimibe versus placebo on the progression of atherosclerosis in the carotid arteries will be assessed using standard ultrasound techniques.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of heterozygous familial hypercholesterolemia
* Ambulatory male (40 to 75 years, inclusive) or female (45 to 75 years, inclusive) subjects
* Calculated LDL-C level greater than or equal to 100 mg/dL (or 2.5 mmol/L) and triglycerides less than 500 mg/dL (5.65 mmol/L) while on usual and stable lipid-lowering therapy

Exclusion Criteria:

* Breast feeding or lactating women
* Previous organ transplantation
* High-grade stenosis (>75%) or the occlusion of any segment of either carotid artery
* History of carotid endarterectomy, or insertion of carotid artery stent or are scheduled to have either of these procedures

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 796
Dates: Start 2004-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To demonstrate the effect of pactimibe versus placebo, when added to usual medical care, on the intima-media thickness (IMT) of the carotid arteries in subjects with heterozygous familial hypercholesterolemia (HeFH) and carotid atherosclerosis.

SECONDARY OUTCOMES:
To assess the effects of pactimibe versus placebo, when added to usual medical care:
- on the incidence and the time to first occurrence of
cardiovascular events,
- on inflammatory and oxidative markers, such as serum
high-sensitivity C-reactive protein (hsCRP), plasma
interleukin 6 (IL-6), plasma myeloperoxidase (MPO) and
serum nitrotyrosine.
To compare the safety of pactimibe versus placebo, when added to usual medical care, particularly with respect to the incidence of clincal and laboratory adverse events.

CONTACTS AND LOCATIONS:
Locations (37):
- United States (8):
  - Santa Ana, California
  - Chicago, Illinois
  - Baltimore, Maryland
  - St Louis, Missouri
  - Cincinnati, Ohio
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- Canada (6):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Chomedey Laval, Quebec
  - Montreal, Quebec
  - Ste-Foy, Quebec
- Jerusalem, Israel
- Netherlands (12):
  - Amsterdam, Zuidoost
  - Capelle aan den IJssel
  - Dordrecht
  - Etten-Leur
  - Goes
  - Gorinchem
  - Gouda
  - Groningen
  - Hoorn
  - Leiden
  - Rotterdam
  - Tilburg
- Oslo, Norway
- South Africa (3):
  - Bellville
  - Midrand
  - Pretoria
- Spain (2):
  - Barcelona
  - Córdoba
- Sweden (2):
  - Linköping
  - Stockholm
- United Kingdom (2):
  - London
  - Manchester

REFERENCES:
- [Derived] Meuwese MC, de Groot E, Duivenvoorden R, Trip MD, Ose L, Maritz FJ, Basart DC, Kastelein JJ, Habib R, Davidson MH, Zwinderman AH, Schwocho LR, Stein EA; CAPTIVATE Investigators. ACAT inhibition and progression of carotid atherosclerosis in patients with familial hypercholesterolemia: the CAPTIVATE randomized trial. JAMA. 2009 Mar 18;301(11):1131-9. doi: 10.1001/jama.301.11.1131. PMID 19293413